CLINICAL TRIAL: NCT03169439
Title: Irreversible Electroporation for Treatment of Solid Abdominal Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Jolie Welson, principle investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IREAT
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hepatic focal lesions and pancreatic masses (Other)
  Interventions: Procedure: Irreversible electroporation

INTERVENTIONS:
Procedure: Irreversible electroporation — minimal invasive ablative technique for tumors

SUMMARY:
Irreversible electroporation (IRE) is a novel non-thermal ablation modality with promise for revolutionizing the treatment for local solid tumors.

With the growing demand for alternative and less invasive treatments for localized tumors, the investigators have seen the development and investigation of several tissue ablation modalities, including radiofrequency ablation (RFA), microwave ablation, and cryoablation. Although these modalities have been efficacious, they have some disadvantages owing to their reliance on thermal energy for creating cell death.

DETAILED DESCRIPTION:
Irreversible electroporation is novel in that it does not use thermal energy, but electrical energy to produce focused cell death while sparing the normal extracellular matrix, nearby vessels, and structures, while allowing for rapid normal tissue regrowth.

Unlike thermal ablation modalities, Irreversible electroporation does not require significant consideration for dissipation of thermal energy, or heat sink, and has less complications relating to damage of normal soft tissue, eliminating a major cause of treatment failure.

Irreversible electroporation is a novel minimally invasive tumor/tissue ablation technique that can be used under guidance of ultrasound (US) or computed tomography (CT), without inducing thermal damaging effects, and with preservation of the surrounding vital structures such as vessels, bile ducts, urethra, and nerves which remain intact to function normally, even in locally advanced tumors. The technique depends upon inducing apoptotic non-necrotic cell death in short procedure time.

It has the advantage of allowing quick tissue regeneration. Irreversible electroporation treatment time is significantly shorter than traditional thermal ablation modalities, usually in few minutes range, and allows for treating considerably larger lesions than thermal ablation modalities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable solid abdominal tumors (hepatic, pancreatic, porta hepatis,…).
* The mass measures less than 4 cm.
* Associated with no or oligo metastatic lesions

Exclusion Criteria:

* Patients with cardiac arrhythmia and pacemaker.
* Patients unfit for general anesthesia.
* The lesion size is larger than 4 cm.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
The ablation success | 3 months
  the ability to deliver planned therapy and to have no residual

SECONDARY OUTCOMES:
Local recurrence | 3,6 and 12 months
  defined as re appearance of viable tumor after period during which no tumor could be detected

REFERENCES:
- [Background] Davalos RV, Mir IL, Rubinsky B. Tissue ablation with irreversible electroporation. Ann Biomed Eng. 2005 Feb;33(2):223-31. doi: 10.1007/s10439-005-8981-8. PMID 15771276
- [Background] Edd JF, Horowitz L, Davalos RV, Mir LM, Rubinsky B. In vivo results of a new focal tissue ablation technique: irreversible electroporation. IEEE Trans Biomed Eng. 2006 Jul;53(7):1409-15. doi: 10.1109/TBME.2006.873745. PMID 16830945
- [Background] Lee EW, Chen C, Prieto VE, Dry SM, Loh CT, Kee ST. Advanced hepatic ablation technique for creating complete cell death: irreversible electroporation. Radiology. 2010 May;255(2):426-33. doi: 10.1148/radiol.10090337. PMID 20413755
- [Background] Rubinsky B. Irreversible electroporation in medicine. Technol Cancer Res Treat. 2007 Aug;6(4):255-60. doi: 10.1177/153303460700600401. PMID 17668932
- [Background] Kasivisvanathan V, Thapar A, Oskrochi Y, Picard J, Leen EL. Irreversible electroporation for focal ablation at the porta hepatis. Cardiovasc Intervent Radiol. 2012 Dec;35(6):1531-4. doi: 10.1007/s00270-012-0363-7. Epub 2012 Feb 25. PMID 22367010
- [Background] Usman M, Moore W, Talati R, Watkins K, Bilfinger TV. Irreversible electroporation of lung neoplasm: a case series. Med Sci Monit. 2012 Jun;18(6):CS43-7. doi: 10.12659/msm.882888. PMID 22648257
- [Background] Esser AT, Smith KC, Gowrishankar TR, Weaver JC. Towards solid tumor treatment by nanosecond pulsed electric fields. Technol Cancer Res Treat. 2009 Aug;8(4):289-306. doi: 10.1177/153303460900800406. PMID 19645522
- [Background] Silk MT, Wimmer T, Lee KS, Srimathveeravalli G, Brown KT, Kingham PT, Fong Y, Durack JC, Sofocleous CT, Solomon SB. Percutaneous ablation of peribiliary tumors with irreversible electroporation. J Vasc Interv Radiol. 2014 Jan;25(1):112-8. doi: 10.1016/j.jvir.2013.10.012. Epub 2013 Nov 18. PMID 24262034